CLINICAL TRIAL: NCT06171399
Title: The Impact of Cannabis Edibles Packaging Descriptors on Consumer Appeal, Harm Perceptions and Willingness to Try
Brief Title: Cannabis Edibles Packaging Descriptors Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00104038; R01DA053209 (NIH)
Record Dates: First submitted 2023-12-05; First posted 2023-12-14 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2023-11

CONDITIONS: Cannabis Use
Keywords: Cannabis use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- "All Natural" descriptor (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with the product descriptor "All Natural."
  Interventions: Behavioral: "All Natural" descriptor
- "Gluten-free" descriptor (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with the product descriptor "Gluten-free"
  Interventions: Behavioral: "Gluten-free" descriptor
- "Vegan" descriptor (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with the product descriptor "Vegan"
  Interventions: Behavioral: "Vegan" descriptor
- "100% Organic" descriptor (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with the product descriptor "100% Organic"
  Interventions: Behavioral: "100% Organic" descriptor
- "Handcrafted" descriptor (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with the product descriptor "Handcrafted"
  Interventions: Behavioral: "Handcrafted" descriptor
- "Made with live resin" descriptor (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with the product descriptor "Made with live resin"
  Interventions: Behavioral: "Made with live resin" descriptor
- "Fast-acting" descriptor (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with the product descriptor "Fast-acting"
  Interventions: Behavioral: "Fast-acting" descriptor
- "Relax" descriptor (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with the product descriptor "Relax"
  Interventions: Behavioral: "Relax" descriptor
- "Energy Boost" descriptor (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) with the product descriptor "Energy Boost"
  Interventions: Behavioral: "Energy Boost" descriptor
- No descriptor (control) (Experimental): Four edible product packages (gummies, chocolate, mints, cookies) without any product descriptors
  Interventions: Behavioral: No descriptor (control)

INTERVENTIONS:
Behavioral: "All Natural" descriptor — Participants in the nine intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the product descriptors of interest. All participants will see the same four products, and each condition will see the products with the same descriptor.
  Arms: "All Natural" descriptor
Behavioral: "Gluten-free" descriptor — Participants in the nine intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the product descriptors of interest. All participants will see the same four products, and each condition will see the products with the same descriptor.
  Arms: "Gluten-free" descriptor
Behavioral: "Vegan" descriptor — Participants in the nine intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the product descriptors of interest. All participants will see the same four products, and each condition will see the products with the same descriptor.
  Arms: "Vegan" descriptor
Behavioral: "100% Organic" descriptor — Participants in the nine intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the product descriptors of interest. All participants will see the same four products, and each condition will see the products with the same descriptor.
  Arms: "100% Organic" descriptor
Behavioral: "Handcrafted" descriptor — Participants in the nine intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the product descriptors of interest. All participants will see the same four products, and each condition will see the products with the same descriptor.
  Arms: "Handcrafted" descriptor
Behavioral: "Made with live resin" descriptor — Participants in the nine intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the product descriptors of interest. All participants will see the same four products, and each condition will see the products with the same descriptor.
  Arms: "Made with live resin" descriptor
Behavioral: "Fast-acting" descriptor — Participants in the nine intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the product descriptors of interest. All participants will see the same four products, and each condition will see the products with the same descriptor.
  Arms: "Fast-acting" descriptor
Behavioral: "Relax" descriptor — Participants in the nine intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the product descriptors of interest. All participants will see the same four products, and each condition will see the products with the same descriptor.
  Arms: "Relax" descriptor
Behavioral: "Energy Boost" descriptor — Participants in the nine intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the product descriptors of interest. All participants will see the same four products, and each condition will see the products with the same descriptor.
  Arms: "Energy Boost" descriptor
Behavioral: No descriptor (control) — Participants in the nine intervention conditions will be shown four cannabis edibles packages that have been altered to contain one of the product descriptors of interest. All participants will see the same four products, and each condition will see the products with the same descriptor.
  Arms: No descriptor (control)

SUMMARY:
The purpose of this study is to assess differences in perceptions of product appeal, harm, and subsequent willingness to try cannabis edibles products with/without product descriptors of interest.

DETAILED DESCRIPTION:
Cannabis edibles are rapidly leading the legal recreational cannabis market. They present health harms that are not typical of smoked marijuana, including accidental overconsumption of high levels of Delta-9-tetrahydrocannabinol (THC). Product packaging plays an important role in influencing perceptions of a product's appeal and potential harm. This experiment will assign participants to view real cannabis edibles packaging edited with one of nine commonly used product descriptors found on real cannabis edibles products, and ask a series of questions to assess perceptions of product appeal and harm. One group of participants will serve as the control and will see the same cannabis edibles packaging without any product descriptors.

ELIGIBILITY:
Inclusion Criteria:

* US resident
* Aged 18-65, inclusive
* Up to 13% of participants will be those who identify as Black/African American
* Up to 16% of participants will be those who identify as Hispanic
* Approximately 50% of participants will be past year cannabis users

Exclusion Criteria:

* Does not currently reside in the United States
* Younger than 18 or older than 65
* Does not provide information regarding history of cannabis use
* Otherwise eligible but demographic and/or user group quotas have been met

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2521 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Reboussin, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant were recruited from a collection of online survey panels.
Period: Overall Study
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor
Started | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248
Completed | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor | Total
Number analyzed (Participants) | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248 | 2521
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (13.5) | 40.5 (12.9) | 42.6 (13.5) | 41.5 (13.7) | 42.3 (13.2) | 41.6 (13.2) | 41.3 (12.8) | 41.4 (13.4) | 40.8 (13.8) | 42.0 (13.1) | 41.5 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 144 | 135 | 136 | 135 | 132 | 129 | 130 | 126 | 123 | 1310
  Male | 129 | 111 | 117 | 123 | 121 | 121 | 138 | 103 | 123 | 125 | 1211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 56 | 63 | 60 | 69 | 60 | 73 | 55 | 59 | 68 | 619
  Not Hispanic or Latino | 193 | 199 | 189 | 199 | 187 | 193 | 194 | 178 | 190 | 180 | 1902
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 8 | 7 | 4 | 6 | 4 | 2 | 6 | 4 | 48
  Asian | 6 | 4 | 9 | 14 | 8 | 9 | 11 | 11 | 5 | 7 | 84
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 1 | 4 | 1 | 14
  Black or African American | 46 | 64 | 47 | 51 | 55 | 56 | 57 | 51 | 42 | 44 | 513
  White | 168 | 161 | 158 | 152 | 158 | 157 | 164 | 143 | 167 | 160 | 1588
  More than one race | 12 | 13 | 11 | 12 | 12 | 11 | 15 | 12 | 7 | 11 | 116
  Unknown or Not Reported | 12 | 9 | 16 | 22 | 18 | 13 | 16 | 13 | 18 | 21 | 158
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248 | 2521

OUTCOME MEASURES:

1. Primary Outcome: Product Appeal
Description: One item to assess the appeal of the product. Results will be reported as mean for all products within condition. Question: How appealing is this product to you? Response Options: (0) Not at all appealing to (10) Very appealing
Time Frame: After exposure to product packaging up to 1 minute
Measure: Mean (Standard Error); unit: score on a scale 0-10
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor
Number analyzed (Participants) | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248
score on a scale 0-10 | 6.43 (0.17) | 6.04 (0.17) | 6.04 (0.18) | 6.06 (0.17) | 5.73 (0.19) | 6.29 (0.17) | 6.18 (0.17) | 6.10 (0.19) | 6.15 (0.17) | 6.02 (0.18)

2. Primary Outcome: Product Harm Perceptions (Absolute)
Description: One item to assess participants' opinions of safety of the product. Results will be reported as the number of each type of response. Question: How safe do you think it would be to eat the edible in this package? Response options: (1) Completely unsafe, (2) Somewhat unsafe, (3) Somewhat safe, (4) Completely safe
Time Frame: After exposure to product packaging up to 1 minute
Population: Each participant was asked the same question for all four cannabis products shown in their condition. The outcome is the number of responses for all questions for all products within condition.
Measure: Count of Units; unit: Responses per condition
Units Other Than Participants: Responses per condition
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor
Number analyzed (Participants) | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248
Number analyzed (Responses per condition) | 995 | 1018 | 1007 | 1035 | 1024 | 1012 | 1064 | 931 | 994 | 992
Responses per condition
  (1) Completely unsafe | 53 | 67 | 81 | 65 | 95 | 75 | 99 | 80 | 39 | 95
  (2) Somewhat unsafe | 91 | 103 | 94 | 118 | 91 | 77 | 89 | 105 | 115 | 83
  (3) Somewhat safe | 436 | 453 | 452 | 463 | 425 | 517 | 514 | 407 | 484 | 417
  (4) Completely safe | 415 | 395 | 380 | 389 | 413 | 343 | 362 | 339 | 356 | 397

3. Primary Outcome: Willingness to Try Free Sample
Description: One item to assess participants' willingness to try a free sample of the product shown. Results will be reported as the number of each type of response. Question: How interested would you be in a free sample of this product? Response Options: (1) Not at all; (2) Slightly; (3) Somewhat; (4) Moderately; (5) Very
Time Frame: After exposure to product packaging up to 1 minute
Population: as for outcome 2
Measure: Count of Units; unit: Responses per condition
Units Other Than Participants: Responses per condition
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor
Number analyzed (Participants) | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248
Number analyzed (Responses per condition) | 996 | 1020 | 1008 | 1036 | 1024 | 1011 | 1068 | 931 | 996 | 991
Responses per condition
  (1) Not at all | 168 | 215 | 210 | 193 | 234 | 190 | 220 | 198 | 177 | 194
  (2) Slightly | 67 | 83 | 97 | 81 | 88 | 80 | 81 | 72 | 99 | 97
  (3) Somewhat | 140 | 149 | 139 | 169 | 147 | 164 | 146 | 124 | 169 | 143
  (4) Moderately | 188 | 197 | 176 | 201 | 188 | 193 | 206 | 179 | 168 | 171
  (5) Very | 433 | 376 | 386 | 392 | 367 | 384 | 415 | 358 | 383 | 386

4. Primary Outcome: Package Appeal
Description: One item to assess appeal of the packaging of the product. Results with be reported as mean for all products within conditions. Question: How appealing is this packaging to you? Response Options: (0) Not at all appealing to (10) Very appealing
Time Frame: 1 min
Measure: Mean (Standard Error); unit: Score on a scale 0-10
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor
Number analyzed (Participants) | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248
Score on a scale 0-10 | 6.71 (0.15) | 6.28 (0.16) | 6.34 (0.17) | 6.30 (0.16) | 6.11 (0.18) | 6.56 (0.15) | 6.49 (0.16) | 6.41 (0.18) | 6.34 (0.16) | 6.27 (0.17)

5. Primary Outcome: Package Harm Perceptions (Absolute)
Description: One item to assess participants' opinions of product safety based on the packaging. Results will be reported as the number of each type of response. Question: How much does this packaging make you think this edible is safe to consume? Response Options: (1) Not at all; (2) A little; (3) Somewhat; (4) A lot
Time Frame: After exposure to product packaging up to 1 min
Population: as for outcome 2
Measure: Count of Units; unit: Responses per condition
Units Other Than Participants: Responses per condition
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor
Number analyzed (Participants) | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248
Number analyzed (Responses per condition) | 994 | 1019 | 1007 | 1035 | 1023 | 1010 | 1067 | 931 | 994 | 991
Responses per condition
  (1) Not at all | 85 | 110 | 122 | 101 | 123 | 109 | 130 | 126 | 93 | 122
  (2) A little | 145 | 139 | 171 | 188 | 169 | 186 | 165 | 167 | 188 | 177
  (3) Somewhat | 406 | 442 | 380 | 423 | 387 | 438 | 444 | 353 | 392 | 342
  (4) A lote | 358 | 328 | 334 | 323 | 344 | 277 | 328 | 285 | 321 | 350

6. Primary Outcome: Willingness to Try Product
Description: One item to assess the participants' willingness to try the product based on the packaging. Results will be reported as the number of each type of response. Question: How much does seeing this packaging make you want to try this edible? Response Options: (1) Not at all; (2) A little; (3) Somewhat; (4) A lot
Time Frame: After exposure to product packaging up to 1 min
Population: as for outcome 2
Measure: Count of Units; unit: Responses per condition
Units Other Than Participants: Responses per condition
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor
Number analyzed (Participants) | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248
Number analyzed (Responses per condition) | 994 | 1019 | 1007 | 1033 | 1024 | 1011 | 1066 | 930 | 995 | 990
Responses per condition
  (1) Not at all | 171 | 209 | 230 | 217 | 229 | 207 | 213 | 204 | 187 | 204
  (2) A little | 154 | 180 | 185 | 162 | 196 | 172 | 175 | 152 | 183 | 175
  (3) Somewhat | 297 | 324 | 272 | 330 | 284 | 328 | 336 | 257 | 307 | 280
  (4) A lot | 372 | 306 | 320 | 324 | 315 | 304 | 342 | 317 | 318 | 331

7. Secondary Outcome: Appeal to Children Responses
Description: One item to assess the participants' assessment of the product packaging's potential appeal to children. Results will be reported as mean for all products within condition. Questions: How appealing do you think this packaging would be to children? Response Options: (0) Not at all appealing to (10) Very appealing
Time Frame: After exposure to product packaging up to 1 minute
Measure: Mean (Standard Error); unit: Scores on a scale 0-10
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor
Number analyzed (Participants) | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248
Scores on a scale 0-10 | 5.97 (0.15) | 5.71 (0.15) | 5.58 (0.17) | 5.58 (0.16) | 5.34 (0.17) | 5.87 (0.16) | 5.61 (0.16) | 5.84 (0.17) | 5.67 (0.17) | 5.57 (0.18)

8. Secondary Outcome: Product Harm Perceptions (Relative)
Description: One question assessing participants' opinions of safety of the product compared to other, similar, products. Results will be reported as the number of each type of response. Question: Compared to other edible products on the market, how safe do you think the edible in this package is? Response Options: (1) Much less safe; (2) Somewhat less safe; (3) As safe; (4) Somewhat safer; (5) Much safer
Time Frame: After exposure to product packaging up to 1 minute
Population: as for outcome 2
Measure: Count of Units; unit: Responses per condition
Units Other Than Participants: Responses per condition
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor
Number analyzed (Participants) | 249 | 255 | 252 | 259 | 256 | 253 | 267 | 233 | 249 | 248
Number analyzed (Responses per condition) | 996 | 1020 | 1008 | 1036 | 1024 | 1011 | 1068 | 930 | 995 | 991
Responses per condition
  (1) Much less safe | 44 | 48 | 63 | 61 | 82 | 53 | 74 | 70 | 34 | 88
  (2) Somewhat less safe | 52 | 71 | 59 | 70 | 70 | 58 | 66 | 51 | 74 | 59
  (3) As safe | 490 | 486 | 478 | 479 | 464 | 522 | 533 | 422 | 520 | 456
  (4) Somewhat safer | 215 | 246 | 203 | 225 | 220 | 217 | 219 | 206 | 188 | 214
  (5) Much safer | 195 | 169 | 205 | 201 | 188 | 161 | 176 | 181 | 179 | 174

9. Other Pre Specified Outcome: Perception of Quality
Description: One item to assess the participants' perceptions of the quality of the product. Results will be reported as the number of each type of response. Question: To what extent do you agree or disagree that this looks like a good quality product? Response options: (1) Strongly disagree to (5) Strongly agree
Time Frame: After exposure to product packaging up to 1 minute
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Perception of Good Taste
Description: One item to assess the participants' perceptions of the taste of the product. Results will be reported as the number of each type of response. Question: To what extent do you agree or disagree that this edible might taste good? Response options: (1) Strongly disagree to (5) Strongly agree
Time Frame: After exposure to product packaging up to 1 min
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Perception of Healthfulness of Product
Description: One item to asses the participants' perceptions of the healthfulness of the product based on the packaging. Results will be reported as the number of each type of response. Question: How much does this packaging make you think this edible is healthy? Response options: (1) Not at all; (2) A little; (3) Somewhat; (4) A lot
Time Frame: After exposure to product packaging up to 1 min
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 minute
Arm/Group | No Descriptor (Control) | "All Natural" Descriptor | "100% Organic" Descriptor | "Gluten-free" Descriptor | "Vegan" Descriptor | "Handcrafted" Descriptor | "Energy Boost" Descriptor | "Relax" Descriptor | "Fast-acting" Descriptor | "Made With Live Resin" Descriptor
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/255 | 0/252 | 0/259 | 0/256 | 0/253 | 0/267 | 0/233 | 0/249 | 0/248
Serious Adverse Events (participants affected / at risk) | 0/249 | 0/255 | 0/252 | 0/259 | 0/256 | 0/253 | 0/267 | 0/233 | 0/249 | 0/248
Other Adverse Events (participants affected / at risk) | 0/249 | 0/255 | 0/252 | 0/259 | 0/256 | 0/253 | 0/267 | 0/233 | 0/249 | 0/248

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT06171399/Prot_SAP_001.pdf
  • Informed Consent Form (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT06171399/ICF_002.pdf